CLINICAL TRIAL: NCT03735667
Title: ACURATE IDE: Transcatheter Replacement of Stenotic Aortic Valve Through Implantation of ACURATE in Subjects InDicatEd for TAVR
Brief Title: ACURATE IDE: Safety and Effectiveness Study of ACURATE Valve for Transcatheter Aortic Valve Replacement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2408
Record Dates: First submitted 2018-11-06; First posted 2018-11-08 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (7):
- ACURATE Valve - Main Randomized (Experimental): Patients assigned to this group will be implanted with ACURATE neo2™ transfemoral TAVR System.
  *A subset of subjects will also be enrolled in the 4D CT Imaging Substudy.
  Interventions: Device: ACURATE neo2™ Transfemoral TAVR System
- ACURATE Valve - Single-arm Roll-in (Experimental): Patients assigned to this group will be implanted with ACURATE neo2™ transfemoral TAVR System.
  Interventions: Device: ACURATE neo2™ Transfemoral TAVR System
- Commercial Valve - Main Randomized (Active Comparator): Medtronic CoreValve TAVR System OR, Edwards SAPIEN 3 TAVR System
  Patients assigned to this group will be implanted with commercially available balloon-expandable SAPIEN 3™ Transcatheter Heart Valve or future iteration (SAPIEN 3; Edwards Lifesciences LLC, Irvine, CA, USA) or a commercially available self-expanding CoreValve® Transcatheter Aortic Valve Replacement System, CoreValve® Evolut™ R Recapturable TAVR System, EVOLUT™ PRO System, or future iteration (CoreValve; Medtronic, Inc., Dublin, Ireland) TAVR device.
  *A minimum of 200 subjects will also be enrolled in the 4D CT Imaging Substudy.
  Interventions: Device: Medtronic CoreValve TAVR System; Device: Edwards SAPIEN 3 TAVR System
- ACURATE Valve - Single-arm Prime XL (Experimental): Patients assigned to this group will be implanted with ACURATE Prime™ transfemoral TAVR System XL.
  *50 subjects will be enrolled in the Prime™ XL Nested Registry
  Interventions: Device: ACURATE Prime™ Transfemoral TAVR System XL
- ACURATE Valve - Extended Durability Randomized (Experimental): Patients assigned to this group will be implanted with ACURATE neo2™ transfemoral TAVR System (S, M, L) or ACURATE Prime™ transfemoral TAVR System XL. Only low risk patients are enrolled in this group.
  Interventions: Device: ACURATE neo2™ Transfemoral TAVR System; Device: ACURATE Prime™ Transfemoral TAVR System XL
- Commercial Valve - Extended Durability Randomized (Active Comparator): Medtronic CoreValve TAVR System OR, Edwards SAPIEN 3 TAVR System
  Patients assigned to this group will be implanted with commercially available balloon-expandable SAPIEN 3™ Transcatheter Heart Valve or future iteration (SAPIEN 3; Edwards Lifesciences LLC, Irvine, CA, USA) or a commercially available self-expanding CoreValve® Transcatheter Aortic Valve Replacement System, CoreValve® Evolut™ R Recapturable TAVR System, EVOLUT™ PRO System, or future iteration (CoreValve; Medtronic, Inc., Dublin, Ireland) TAVR device. Only low risk patients are enrolled in this group.
  Interventions: Device: Medtronic CoreValve TAVR System; Device: Edwards SAPIEN 3 TAVR System
- ACURATE Valve - Continued Access Study (Experimental): Patients assigned to this group will be implanted with ACURATE neo2™ transfemoral TAVR System (S, M, L) or ACURATE Prime™ transfemoral TAVR System XL.
  Interventions: Device: ACURATE neo2™ Transfemoral TAVR System; Device: ACURATE Prime™ Transfemoral TAVR System XL

INTERVENTIONS:
Device: ACURATE neo2™ Transfemoral TAVR System — ACURATE neo2™ Transfemoral TAVR system: Support frame made of nitinol, supra-annular processed tri-leaflet porcine pericardial valve and an outer skirt to limit paravalvular regurgitation (manufactured by Boston Scientific Corporation, Marlborough, MA, USA).
  Arms: ACURATE Valve - Continued Access Study; ACURATE Valve - Extended Durability Randomized; ACURATE Valve - Main Randomized; ACURATE Valve - Single-arm Roll-in
Device: Medtronic CoreValve TAVR System — Medtronic CoreValve Evolut R or Evolut PRO Transcatheter Aortic Valve Replacement (TAVR) System (or any future Corevalve iterations): The support frame is manufactured from nitinol, which has multilevel, self-expanding properties and is radiopaque. The bioprosthesis is manufactured by suturing valve leaflets and a skirt from porcine pericardium into a tri-leaflet configuration (manufactured by Medtronic CoreValve LLC, Santa Ana, USA).
  Arms: Commercial Valve - Extended Durability Randomized; Commercial Valve - Main Randomized
Device: Edwards SAPIEN 3 TAVR System — Edwards SAPIEN 3 TAVR system (or any future SAPIEN iterations): balloon-expandable transcatheter aortic bioprosthesis, support frame made of cobalt-chromium, three leaflets constructed of processed bovine pericardial tissue and an outer polyethylene terephthalate (PET) sealing cuff to mitigate paravalvular regurgitation (manufactured by Edwards Lifesciences, Inc., Irvine, California, USA)
  Arms: Commercial Valve - Extended Durability Randomized; Commercial Valve - Main Randomized
Device: ACURATE Prime™ Transfemoral TAVR System XL — ACURATE Prime™ Transfemoral TAVR system: Support frame made of nitinol, supra-annular processed tri-leaflet porcine pericardial valve and an outer skirt to limit paravalvular regurgitation (manufactured by Boston Scientific Corporation, Marlborough, MA, USA).
  Arms: ACURATE Valve - Continued Access Study; ACURATE Valve - Extended Durability Randomized; ACURATE Valve - Single-arm Prime XL

SUMMARY:
To evaluate safety and effectiveness of the ACURATE Transfemoral Aortic Valve System for transcatheter aortic valve replacement (TAVR) in subjects with severe native aortic stenosis who are indicated for TAVR.

As of 28-May-2025, Boston Scientific Corporation (BSC) announced the voluntary global discontinuation of the ACURATE product platform, including both the ACURATE neo2 and ACURATE Prime Aortic Valve Systems. BSC will no longer pursue regulatory approval for the device in the U.S. or other unapproved geographies.

DETAILED DESCRIPTION:
Subjects will be enrolled at up to 85 centers in the United States, Canada, Europe, and Australia. There will be up to 2,820 subjects in ACURATE IDE.

The ACURATE IDE study cohorts include the following.

* Main Randomized Cohort: A prospective, multicenter, 1:1 randomized controlled trial (RCT; ACURATE versus a commercially available balloon-expandable SAPIEN 3™ Transcatheter Heart Valve or future iteration [SAPIEN 3; Edwards Lifesciences LLC, Irvine, CA, USA] or a commercially available self-expanding CoreValve® Transcatheter Aortic Valve Replacement System, CoreValve® Evolut™ R Recapturable TAVR System, EVOLUT™ PRO System, or future iteration [CoreValve; Medtronic, Inc., Dublin, Ireland]). There will be up to 1,500 subjects in the RCT.
* Roll-In Cohort: A non-randomized roll-in phase with the test device. Centers that do not have implantation experience with the ACURATE neo™ Aortic Bioprosthesis (transfemoral delivery; Boston Scientific Corporation, Marlborough, MA, USA) will perform at least 2 roll-in cases before commencing treatment in the randomized cohort. Centers with prior experience with ACURATE are not required to do roll-in cases. Data from roll-in subjects will be summarized separately from the randomized cohort and will not be included in the primary endpoint analysis.
* 4D CT Imaging Substudy: Selected centers with the ability to perform high quality 4D computer tomography (CT) scans will include subjects in a 4D CT Imaging Substudy to assess the prevalence of reduced leaflet mobility and hypoattenuated leaflet thickening (HALT) and the relationship, if any, to clinical events. Subjects will be randomized to test (ACURATE) and control device.
* ACURATE Prime™ XL Nested Registry: A non-randomized, nested registry cohort of subjects who will receive the ACURATE Prime™ Transfemoral Aortic Valve System XL (ACURATE Prime XL Nested Registry). Participating centers will be a subset of United States centers that have enrolled subjects in ACURATE IDE. Data from subjects in this nested registry will be summarized separately from the randomized and roll-in cohorts.
* ACURATE Extended Durability Study: An additional 1:1 randomized study (ACURATE versus a commercially available balloon-expandable SAPIEN 3™ Transcatheter Heart Valve or future iteration [SAPIEN 3; Edwards Lifesciences LLC, Irvine, CA, USA] or a commercially available self-expanding CoreValve® Transcatheter Aortic Valve Replacement System, CoreValve® Evolut™ R Recapturable TAVR System, EVOLUT™ PRO System, or future iteration [CoreValve; Medtronic, Inc., Dublin, Ireland]) including only subjects considered to be at low surgical risk. Subjects will receive ACURATE neo2 (S, M, or L valve sizes) or ACURATE Prime XL. Data from subjects in the Extended Durability Study will be summarized separately from other cohorts.
* ACURATE Continued Access Study (CAS): An additional cohort of subjects receiving ACURATE neo2 (S, M, and L valve sizes) or ACURATE Prime XL. Data from subjects in the ACURATE CAS will be summarized separately from other cohorts and will be used to further assess performance and safety.

Follow-up

* Subjects implanted with a test device will be assessed at baseline, peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, 1 year, and then annually for 5 years post-procedure.
* Subjects implanted with a control device will be assessed at baseline, peri- and post-procedure, at discharge or 7 days post procedure (whichever comes first), 30 days, 6 months, and 1 year post procedure. Per protocol, no additional follow-up is required beyond this period, and standard of care practices will apply.
* Some subjects may have completed additional annual follow-up visits based on requirements outlined in earlier versions of the protocol.
* Subjects who are enrolled but not implanted with a test or control device at the time of the procedure will be followed for safety through 1 year.

ELIGIBILITY:
Inclusion Criteria:

* IC1. Subject has documented severe symptomatic native aortic stenosis defined as follows: aortic valve area (AVA) ≤1.0 cm2 (or AVA index ≤0.6 cm2/m2) AND a mean pressure gradient ≥40 mmHg, OR maximal aortic valve velocity ≥4.0 m/s, OR Doppler velocity index ≤0.25 as measured by echocardiography and/or invasive hemodynamics.

Note: In cases of low flow, low gradient aortic stenosis with left ventricular dysfunction (ejection fraction <50%), dobutamine can be used to assess the grade of aortic stenosis (maximum dobutamine dose of 20 mcg/kg/min recommended); the subject may be enrolled if echocardiographic criteria are met with this augmentation.

* IC2. Subject has a documented aortic annulus size of ≥20.5 mm and ≤29 mm based on the center's assessment of pre-procedure diagnostic imaging (and confirmed by the Case Review Committee [CRC]) and, for the Main Randomized Cohort and the Extended Durability Study, is deemed treatable with an available size of both test and control device.
* IC3. For subjects with symptomatic aortic valve stenosis per IC1 definition above, functional status is NYHA Functional Class ≥ II.
* IC4. Heart team (which must include an experienced cardiac interventionalist and an experienced cardiac surgeon) agrees that the subject is indicated for TAVR, is likely to benefit from valve replacement, and TAVR is appropriate.
* IC5. Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent.
* IC6. Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.
* IC7. Subject is expected to be able to take the protocol-required adjunctive pharmacologic therapy.

Exclusion Criteria:

* EC1. Subject has a unicuspid or bicuspid aortic valve.
* EC2. Subject has had an acute myocardial infarction within 30 days prior to the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin elevation).
* EC3. Subject has had a cerebrovascular accident or transient ischemic attack clinically confirmed by a neurologist or neuroimaging within the past 6 months prior to study enrollment.
* EC4. Subject is on renal replacement therapy or has eGFR <20.
* EC5. Subject has a pre-existing prosthetic aortic or mitral valve.
* EC6. Subject has severe (4+) aortic, tricuspid, or mitral regurgitation.
* EC7. Subject has moderate or severe mitral stenosis (mitral valve area ≤1.5 cm2 and diastolic pressure half-time ≥150 ms, Stage C or D76).
* EC8. Subject has a need for emergency surgery for any reason.
* EC9. Subject has a history of endocarditis within 6 months of index procedure or evidence of an active systemic infection or sepsis.
* EC10. Subject has echocardiographic evidence of new intra-cardiac vegetation or intraventricular or paravalvular thrombus requiring intervention.
* EC11. Subject has platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.
* EC12. Subject has had a gastrointestinal bleed requiring hospitalization or transfusion within the past 3 months, or has other clinically significant bleeding diathesis or coagulopathy that would preclude treatment with required antiplatelet regimen, or will refuse transfusions.
* EC13. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to the protocol required medications (aspirin, all P2Y12 inhibitors, heparin), or to the individual components of the test or control valve (nickel, titanium, stainless steel, platinum, iridium or polyethylene terephthalate [PET]).
* EC14. Subject has a life expectancy of less than 12 months due to non-cardiac, comorbid conditions based on the assessment of the investigator at the time of enrollment.
* EC15. Subject has hypertrophic cardiomyopathy.
* EC16. Subject has any therapeutic invasive cardiac or vascular procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty, pacemaker implantation, or implantable cardioverter defibrillator implantation, which are allowed).
* EC17. Subject has untreated coronary artery disease, which in the opinion of the treating physician is clinically significant and requires revascularization.
* EC18. Subject has severe left ventricular dysfunction with ejection fraction <20%.
* EC19. Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
* EC20. Subject has arterial access that is not acceptable for the study device (test or control) delivery systems as defined in the device (test or control) Directions For Use.
* EC21. Subject has either of the following:

  * Severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely; marked tortuosity; significant narrowing of the abdominal aorta; severe unfolding of the thoracic aorta; or thick, protruding, ulcerated atheroma in the aortic arch), OR
  * Severe/eccentric calcification of the aortic annulus that would prevent safe implantation of the TAVR prosthesis.
* EC22. Subject has current problems with substance abuse (e.g., alcohol, etc.) that may interfere with the subject's participation in this study.
* EC23. Subject is participating in another investigational drug or device study that has not reached its primary endpoint or subject intends to participate in another investigational device clinical trial within 12 months after index procedure.
* EC24. Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation. Enrollment is permissible after permanent pacemaker implantation.
* EC25. Subject has severe incapacitating dementia.

Additional exclusion criteria apply to subjects considered for enrollment in the CT Imaging Substudy as listed below.

* AEC1. Subject has eGFR <30 mL/min (chronic kidney disease stage IV or stage V)
* AEC2. Subject has atrial fibrillation that cannot be rate controlled to ventricular response rate < 60 bpm.
* AEC3. Subject is expected to undergo chronic anticoagulation therapy after the index procedure.

Note: Subjects treated with short-term anticoagulation post procedure can be included in the CT Imaging Substudy; in these subjects the 30-day imaging will be performed 30 days after discontinuation of anticoagulation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1948 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2029-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Raj R. Makkar, MD, Principal Investigator — Cedars-Sinai Heart Institute; Michael J. Reardon, MD, Principal Investigator — Methodist DeBakey Heart & Vascular Center
Locations (75):
- United States (69):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Good Samaritan, Phoenix, Arizona
  - HonorHealth Scottsdale Healthcare, Scottsdale, Arizona
  - TMC HealthCare, Tucson, Arizona
  - Baptist Health Medical Center, Little Rock, Arkansas
  - Scripps Clinic, La Jolla, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - University of California, Davis Medical Center, Sacramento, California
  - Kaiser Permanente - San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - NorthShore University Health Study Coordinator, Evanston, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - St. John's Hospital (Prairie), Springfield, Illinois
  - St. Vincent's Hospital, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - St. Joseph's Hospital-St. Paul, Saint Paul, Minnesota
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Englewood Health, Englewood, New Jersey
  - Robert Wood Johnson Medical Center, New Brunswick, New Jersey
  - Albany Medical Center, Albany, New York
  - Kaleida Health, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Medical Center/NYPH, New York, New York
  - Cornell Presbyterian - New York, New York, New York
  - Montefiore-Jack D. Weiler Hospital, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Lindner Center for Research and Education at Christ Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Research and Innovation Institute, Columbus, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Providence Heart Institute, Portland, Oregon
  - Sacred Heart Medical Center - Riverbend, Springfield, Oregon
  - UPMC - Pinnacle, Harrisburg, Pennsylvania
  - UPMC Pittsburgh, Pittsburgh, Pennsylvania
  - Lankenau, Wynnewood, Pennsylvania
  - WellSpan York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - St Thomas Ascension, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor Regional Medical Center at Plano, Plano, Texas
  - Methodist Healthcare System of San Antonio dba Methodist Hospital, San Antonio, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Providence Regional Medical Center, Everett, Washington
  - Bellin Health, Green Bay, Wisconsin
  - Aurora Research Institute, Milwaukee, Wisconsin
  - Medical College of Wisconsin - Froedtert Hospital, Milwaukee, Wisconsin
- Canada (6):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Providence Health - St. Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ), Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html)

REFERENCES:
- [Background] Makkar RR, Chakravarty T, Gupta A, Soliman O, Gnall E, Ramana RK, Ramlawi B, Diamantouros P, Potluri S, Kleiman NS, Samy S, Rassi A, Yadav P, Thourani V, Yakubov S, Frawley C, Patel D, Kapadia S, Chalekian A, Modolo R, Sathananthan J, Kim WK, Reardon MJ. Valve Underexpansion and Clinical Outcomes With ACURATE neo2: Findings From the ACURATE IDE Trial. J Am Coll Cardiol. 2025 Jul 29;86(4):225-238. doi: 10.1016/j.jacc.2025.05.011. Epub 2025 May 21. PMID 40406945
- [Result] Makkar RR, Ramana RK, Gnall E, Ramlawi B, Cheng W, Diamantouros P, Potluri S, Kleinman N, Gupta A, Chakravarty T, Samy S, Rassi A, Rajagopal V, Yakubov S, Sorajja P, Patel D, Garcia S, Yadav P, Thourani V, Wang J, Rinaldi M, Kapadia S, Waksman R, Webb J, Ren CB, Gregson J, Modolo R, Sathananthan J, Reardon MJ; ACURATE IDE study investigators. ACURATE neo2 valve versus commercially available transcatheter heart valves in patients with severe aortic stenosis (ACURATE IDE): a multicentre, randomised, controlled, non-inferiority trial. Lancet. 2025 Jun 7;405(10494):2061-2074. doi: 10.1016/S0140-6736(25)00319-8. Epub 2025 May 21. PMID 40412426

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Main Randomized Cohort: 1500 subjects randomized from 10Jun2019 to 19Apr2023. Roll-in Cohort: 148 subjects enrolled from 10Jul2019 to 27Feb2023.
Pre-assignment Details: The non-randomized Roll-in phase with only the test device was for centers with no previous experience implanting ACURATE. Each applicable site performed at least two Roll-in cases before starting enrollment in the Main Randomized Cohort.
  Only data for the Main Randomized Cohort and Roll-in Cohort are being reported at this time as data for the 4D-CT Substudy and other 3 cohorts (Continued Access Study, Extended Durability, and Prime XL Nested Registry) are not available.
Groups:
- ACURATE neo2 Valve - Main Randomized: Patients assigned to this group will be implanted with ACURATE neo2™ transfemoral TAVR System.
  *A subset of subjects will also be enrolled in the 4D CT Imaging Substudy.
- ACURATE neo 2 Valve - Single-arm Roll-in: Patients assigned to this group will be implanted with ACURATE neo2™ transfemoral TAVR System.
Period: 1 Year PE Main Randomized and Roll-in
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo 2 Valve - Single-arm Roll-in
Started | 752 | 748 | 148
Eligible 1-Year | 716 | 720 | 141
Completed | 649 | 658 | 130
Not Completed | 103 | 90 | 18
Not completed — Death | 40 | 31 | 7
Not completed — Lost to Follow-up | 3 | 2 | 0
Not completed — Physician Decision | 4 | 2 | 0
Not completed — Withdrawal by Subject | 27 | 24 | 2
Not completed — 1-Year Visit Not Done | 28 | 29 | 9
Not completed — Other | 1 | 2 | 0
Period: 4D-CT Substudy (subset of Main RCT)
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo 2 Valve - Single-arm Roll-in
Started | 160 | 158 | 0
Eligible 1 Year 4D-CT | 153 | 154 | 0
Completed | 143 | 144 | 0
Not Completed | 17 | 14 | 0
Not completed — Death | 8 | 5 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Other | 0 | 1 | 0
Not completed — 1-Year Visit Not Done | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intention-To-Treat (ITT): This population includes all subjects who sign an Informed Consent Form, are enrolled in the trial, and are randomized, whether or not an assigned study device is implanted. A subject treatment group is based on the randomization assignment.
Groups:
- Commercial Valve - Main Randomized: Medtronic CoreValve TAVR System OR,Edwards SAPIEN 3 TAVR System
  Patients assigned to this group will be implanted with commercially available balloon-expandable SAPIEN 3™ Transcatheter Heart Valve or future iteration (SAPIEN 3; Edwards Lifesciences LLC, Irvine, CA, USA) or a commercially available self-expanding CoreValve® Transcatheter Aortic Valve Replacement System, CoreValve® Evolut™ R Recapturable TAVR System, EVOLUT™ PRO System, or future iteration (CoreValve; Medtronic, Inc., Dublin, Ireland) TAVR device.
  *A minimum of 200 subjects will also be enrolled in the 4D CT Imaging Substudy.
- ACURATE neo2 Valve - Single-arm Roll-in: Patients assigned to this group will be implanted with ACURATE neo2™ transfemoral TAVR System.
- Total: Total of all reporting groups
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in | Total
Number analyzed (Participants) | 752 | 748 | 148 | 1648
Age, Continuous [Mean (Standard Deviation); unit: Years] | 78.0 (6.9) | 79.0 (6.5) | 78.8 (7.1) | 78.5 (6.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 357 | 364 | 64 | 785
  Female | 395 | 383 | 84 | 862
  Intersex | 0 | 0 | 0 | 0
  Unknown | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Note - As subjects had the option to select more than one race/ethnicity, the sum of participants in this Baseline Measure does not equal the overall number of Baseline Participants in each Arm/Group.
  Participants
    American Indian or Alaska Native | 3 | 0 | 1 | 4
    Asian | 6 | 13 | 1 | 20
    Asian - Chinese | 0 | 3 | 0 | 3
    Asian - Japanese | 1 | 0 | 0 | 1
    Asian - Korean | 2 | 1 | 1 | 4
    Other Asian | 3 | 9 | 0 | 12
    Black or African American | 29 | 23 | 3 | 55
    Caucasian | 675 | 659 | 137 | 1471
    Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 1
    Other | 13 | 11 | 2 | 26
    Not Disclosed | 5 | 14 | 1 | 20
    Hispanic or Latino | 24 | 27 | 3 | 54
Region of Enrollment [Number; unit: participants]
  Canada | 59 | 61 | 0 | 120
  United States | 693 | 687 | 148 | 1528
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 30.6 (6.5) | 29.8 (6.1) | 31.5 (7.8) | 30.3 (6.5)
Aortic Annulus Area [Mean (Standard Deviation); unit: mm2] — Computed Tomography Angiography (CTA) Core Laboratory Analysis
  mm2 | 435.2 (58.7) | 437.3 (54.7) | 439.6 (56.6) | 436.5 (56.7)
Aortic Annulus Perimeter [Mean (Standard Deviation); unit: mm] — Computed Tomography Angiography (CTA) Core Laboratory Analysis
  mm | 74.8 (5.0) | 75.1 (4.6) | 75.2 (4.9) | 75.0 (4.8)
Medical History [Number; unit: Percentage of participants]
  History of hypertension | 89.4 | 88.0 | 91.2 | 88.9
  History of coronary artery disease | 52.1 | 52.9 | 58.1 | 53.0
  History of myocardial infarction | 8.6 | 7.8 | 10.8 | 8.4
  History of congestive heart failure | 31.6 | 35.0 | 47.3 | 34.6
  History of atrial fibrillation/atrial flutter | 24.1 | 23.4 | 34.5 | 24.7
  Prior pacemaker implant | 6.4 | 7.0 | 11.5 | 7.1
  History of cerebrovascular accident (TIA & stroke) | 13.0 | 11.5 | 12.2 | 12.3
  Current diabetes mellitus | 37.2 | 36.2 | 42.6 | 37.3
New York Heart Association (NYHA) Classification [Number; unit: Percentage of participants] — NYHA Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  Percentage of participants
    Class I | 0.0 | 0.0 | 0.0 | 0.0
    Class II | 50.7 | 57.8 | 54.7 | 54.2
    Class III | 47.3 | 40.4 | 43.9 | 43.9
    Class IV | 2.0 | 1.9 | 1.4 | 1.9
Operative Risk Group [Number; unit: Percentage of participants] — The subject operative risk is assessed by the site Heart Team and then confirmed by the Case Review Committee who ultimately confirms the subject eligibility for the enrollment in the study.
  Percentage of participants
    High/Extreme | 25.5 | 28.6 | 33.8 | 27.7
    Intermediate | 38.6 | 36.9 | 52.7 | 39.1
    Low | 35.9 | 34.5 | 13.5 | 33.3
Society of Thoracic Surgeons (STS) Risk Score [Mean (Standard Deviation); unit: Percent] — The Society of Thoracic Surgeons Score is a risk model used to predict a subject's risk of mortality and morbidities for the most commonly performed cardiac surgeries. The model is a percentage score from 0 to 100 where a lower score means a lower risk and higher score means a higher risk.
  Percent | 2.7 (1.8) | 2.8 (1.9) | 3.5 (2.3) | 2.8 (1.9)
Aortic Valve Area (AVA) [Mean (Standard Deviation); unit: cm2] — Transthoracic Echocardiography (TTE) - Core Laboratory Analysis Population: Number analyzed participants is based on central echo core lab data. Blank data fields or data recorded in the clinical database as 'Not evaluable' are considered missing.
  cm2
    number analyzed (Participants) | 724 | 716 | 140 | 1580
    (all) | 0.67 (0.14) | 0.67 (0.15) | 0.71 (0.17) | 0.68 (0.15)
Doppler Velocity Index (DVI) [Mean (Standard Deviation); unit: Index] — Transthoracic Echocardiography (TTE) - Core Laboratory Analysis
  DVI=LVOT Velocity/AV Velocity
  * Lower DVI values (< 0.25): Suggest severe aortic stenosis. This indicates that the velocity through the LVOT is much lower relative to the high velocity through the stenotic aortic valve.
  * Intermediate values (approximately 0.25-0.50): May indicate moderate stenosis.
  * Higher DVI values (> 0.50): Are generally considered normal or only mildly abnormal, indicating minimal obstruction. Population: Number analyzed participants is based on central echo core lab data. Blank data fields or data recorded in the clinical database as 'Not evaluable' are considered missing.
  Index
    number analyzed (Participants) | 731 | 718 | 142 | 1591
    (all) | 0.24 (0.05) | 0.24 (0.05) | 0.24 (0.06) | 0.24 (0.05)
Aortic Valve Mean Pressure Gradient [Mean (Standard Deviation); unit: mmHg] — Transthoracic Echocardiography (TTE) - Core Laboratory Analysis Population: Number analyzed participants is based on central echo core lab data. Blank data fields or data recorded in the clinical database as 'Not evaluable' are considered missing.
  mmHg
    number analyzed (Participants) | 734 | 726 | 142 | 1602
    (all) | 39.6 (11.1) | 39.4 (10.5) | 38.7 (12.0) | 39.4 (10.9)
Aortic Valve Peak Velocity [Mean (Standard Deviation); unit: m/s] — Transthoracic Echocardiography (TTE) - Core Laboratory Analysis Population: Number analyzed participants is based on central echo core lab data. Blank data fields or data recorded in the clinical database as 'Not evaluable' are considered missing.
  m/s
    number analyzed (Participants) | 734 | 726 | 142 | 1602
    (all) | 4.05 (0.54) | 4.04 (0.51) | 3.99 (0.57) | 4.04 (0.53)

OUTCOME MEASURES:

1. Primary Outcome: Composite Rate of All-cause Mortality, All Stroke, and Rehospitalization* at 1 Year in the Main Randomized Cohort.
Description: Primary Endpoint: A Clinical Events Committee (CEC), independent group of physician experts reviewed and adjudicated all reported cases of death, stroke and rehospitalization to determine whether they met the specific protocol definition of the event. The CEC adjudicated results are used in the endpoint analysis.
  * Hospitalization for valve-related symptoms or worsening congestive heart failure (NYHA class III or IV); per VARC-2 definition.
Time Frame: Participants will be followed for the duration of hospital stay through 1 year.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized
Number analyzed (Participants) | 752 | 748
percentage of participants | 16.16 [13.38 to 19.07] | 9.53 [7.47 to 11.89]
Statistical Analysis 1: Comparison: ACURATE neo2 Valve - Main Randomized vs Commercial Valve - Main Randomized; Test type: Non-Inferiority — A Bayesian analysis based on 10,000 samples from the posterior distribution, using a piecewise exponential survival model. The criteria for non-inferiority is met if the posterior probability of non-inferiority is greater than the non-inferiority test threshold; A Bayesian analysis was used to test the non-inferiority hypothesis for the primary endpoint using a non-inferiority margin of 8%. The pre-specified success criteria (the non-inferiority test threshold) was a posterior probability of non-inferiority greater than 97.5%. The observed posterior probability of non-inferiority was 77.9%. The posterior median percentage difference in the rate of the primary outcome was 6.63% (95% Bayesian credible interval: 3.04% to 10.20%)

2. Other Pre Specified Outcome: Rate of Mortality: All-cause, Cardiovascular, and Non-cardiovascular
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definition.
Time Frame: Participants will be followed peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 Days, 6 Months, and 1 Year. Data for 2-10 years will be posted once data is complete.
Population: Intention-To-Treat (ITT): This population includes all subjects who sign an ICF, are enrolled in the trial, and are randomized, whether or not an assigned study device is implanted. A subject treatment group is based on the randomization assignment.
  Evaluable for clinical endpoints at 30 days/6 Months/1 Year is defined as subjects who experience an event through 30 days/6 Months/1 Year post-randomization or who were event-free with last follow-up at least 23/150/335 days post- randomization.
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  Mortality: all-cause at Discharge/7 Days Post-Randomization | 0.5 | 0 | 0.7
  Mortality: cardiovascular at Discharge/7 Days Post-Randomization | 0.5 | 0 | 0.7
  Mortality: non-cardiovascular at Discharge/7 Days Post-Randomization | 0 | 0 | 0
  Mortality: all-cause at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Mortality: all-cause at 30 Days Post-Randomization | 0.7 | 0.4 | 1.4
  Mortality: cardiovascular at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Mortality: cardiovascular at 30 Days Post-Randomization | 0.5 | 0.3 | 1.4
  Mortality: non-cardiovascular at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Mortality: non-cardiovascular at 30 Days Post-Randomization | 0.1 | 0.1 | 0
  Mortality: all-cause at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Mortality: all-cause at 6 Months Post-Randomization | 2.7 | 1.2 | 2
  Mortality: cardiovascular at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Mortality: cardiovascular at 6 Months Post-Randomization | 2.1 | 0.5 | 2
  Mortality: non-cardiovascular at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Mortality: non-cardiovascular at 6 Months Post-Randomization | 0.7 | 0.7 | 0
  Mortality: all-cause at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Mortality: all-cause at 1 Year Post-Randomization | 5.0 | 3.9 | 4.8
  Mortality: cardiovascular at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Mortality: cardiovascular at 1 Year Post-Randomization | 3.8 | 1.8 | 3.4
  Mortality: non-cardiovascular at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Mortality: non-cardiovascular at 1 Year Post-Randomization | 1.3 | 2.1 | 1.4

3. Other Pre Specified Outcome: Rate of All Stroke: Disabling and Non-disabling
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definition.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  All stroke at Discharge/7 Days Post-Randomization | 0.9 | 1.1 | 1.4
  Disabling stroke at Discharge/7 Days Post-Randomization | 0.3 | 0.7 | 0.7
  Non-disabling stroke at Discharge/7 Days Post-Randomization | 0.7 | 0.4 | 0.7
  All stroke at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  All stroke at 30 Days Post-Randomization | 1.4 | 1.4 | 1.4
  Disabling stroke at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Disabling stroke at 30 Days Post-Randomization | 0.5 | 0.8 | 0.7
  Non-disabling stroke at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Non-disabling stroke at 30 Days Post-Randomization | 1.0 | 0.5 | 0.7
  All stroke at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  All stroke at 6 Months Post-Randomization | 4.0 | 2.5 | 5.4
  Disabling stroke at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Disabling stroke at 6 Months Post-Randomization | 1.4 | 1.0 | 1.4
  Non-disabling stroke at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Non-disabling stroke at 6 Months Post-Randomization | 2.7 | 1.5 | 4.1
  All stroke at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  All stroke at 1 Year Post-Randomization | 5.7 | 3.5 | 7.5
  Disabling stroke at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Disabling stroke at 1 Year Post-Randomization | 1.9 | 1.3 | 2.1
  Non-disabling stroke at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Non-disabling stroke at 1 Year Post-Randomization | 3.9 | 2.2 | 5.5

4. Other Pre Specified Outcome: Rate of Myocardial Infarction (MI): Periprocedural (≤72 Hours Post Index Procedure) and Spontaneous (>72 Hours Post Index Procedure)
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  MI at Discharge/7 Days Post-Randomization | 0.3 | 0 | 0.7
  Periprocedural MI at Discharge/7 Days Post-Randomization | 0.3 | 0 | 0.7
  Spontaneous MI at Discharge/7 Days Post-Randomization | 0 | 0 | 0
  MI at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  MI at 30 Days Post-Randomization | 0.5 | 0.1 | 0.7
  Periprocedural MI at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Periprocedural MI at 30 Days Post-Randomization | 0.4 | 0 | 0.7
  Spontaneous MI at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Spontaneous MI at 30 Days Post-Randomization | 0.1 | 0.1 | 0
  MI at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  MI at 6 Months Post-Randomization | 1.5 | 0.1 | 0.7
  Periprocedural MI at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Periprocedural MI at 6 Months Post-Randomization | 0.4 | 0 | 0.7
  Spontaneous MI at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Spontaneous MI at 6 Months Post-Randomization | 1.1 | 0.1 | 0
  MI at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  MI at 1 Year Post-Randomization | 2.4 | 0.7 | 0.7
  Periprocedural MI at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Periprocedural MI at 1 Year Post-Randomization | 0.4 | 0 | 0.7
  Spontaneous MI at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Spontaneous MI at 1 Year Post-Randomization | 1.9 | 0.7 | 0

5. Other Pre Specified Outcome: Rate of Bleeding: Life-threatening (or Disabling) and Major
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: Participants will be followed peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 Days, 6 Months, and 1 Year. Data for 2-5 years will be posted once data is complete.
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  Life-threatening or disabling bleeding at Discharge/7 Days Post-Randomization | 1.2 | 1.2 | 2.0
  Major bleeding at Discharge/7 Days Post-Randomization | 1.2 | 1.2 | 0
  Life-threatening or disabling bleeding at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Life-threatening or disabling bleeding at 30 Days Post-Randomization | 1.4 | 1.2 | 2.0
  Major bleeding at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  Major bleeding at 30 Days Post-Randomization | 1.6 | 1.4 | 0.7
  Life-threatening or disabling bleeding at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Life-threatening or disabling bleeding at 6 Months Post-Randomization | 2.9 | 2.3 | 2.0
  Major bleeding at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  Major bleeding at 6 Months Post-Randomization | 2.2 | 2.6 | 2.7
  Life-threatening or disabling bleeding at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Life-threatening or disabling bleeding at 1 Year Post-Randomization | 3.6 | 3.3 | 2.7
  Major bleeding at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  Major bleeding at 1 Year Post-Randomization | 2.9 | 3.3 | 3.4

6. Other Pre Specified Outcome: Rate of Major Vascular Complications
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  Discharge/7 Days Post-Randomization | 2.4 | 1.5 | 1.4
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 2.7 | 1.6 | 1.4
  6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post-Randomization | 3.2 | 2.1 | 2.0
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 3.2 | 2.1 | 2.1

7. Other Pre Specified Outcome: Rate of Repeat Procedure for Valve-related Dysfunction (Surgical or Interventional Therapy)
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  Discharge/7 Days Post-Randomization | 0 | 0 | 0
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 0 | 0 | 0
  6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post-Randomization | 0.1 | 0.1 | 0.7
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 0.1 | 0.4 | 0.7

8. Other Pre Specified Outcome: Rate of Hospitalization for Valve-related Symptoms or Worsening Congestive Heart Failure (NYHA Class III or IV)
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  Discharge/7 Days Post-Randomization | 0 | 0 | 0
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 0.8 | 0.1 | 3.4
  6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post-Randomization | 3.7 | 1.1 | 4.1
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 5.3 | 3.5 | 4.8

9. Other Pre Specified Outcome: Rate of New Permanent Pacemaker Implantation (PPI) Resulting From New or Worsened Conduction Disturbances
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  Discharge/7 Days Post-Randomization | 5.3 | 6.3 | 1.4
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 8.6 | 9.5 | 4.7
  6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post-Randomization | 10.7 | 10.9 | 7.4
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 11.4 | 12.2 | 8.2

10. Other Pre Specified Outcome: Rate of New Onset of Atrial Fibrillation or Atrial Flutter
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  New onset of atrial fibrillation at Discharge/7 Days Post-Randomization | 1.9 | 2.1 | 2.7
  New onset of atrial flutter at Discharge/7 Days Post-Randomization | 0 | 0.1 | 0
  New onset of atrial fibrillation at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  New onset of atrial fibrillation at 30 Days Post-Randomization | 2.2 | 2.2 | 3.4
  New onset of atrial flutter at 30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  New onset of atrial flutter at 30 Days Post-Randomization | 0 | 0.1 | 0
  New onset of atrial fibrillation at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  New onset of atrial fibrillation at 6 Months Post-Randomization | 2.3 | 2.3 | 3.4
  New onset of atrial flutter at 6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  New onset of atrial flutter at 6 Months Post-Randomization | 0 | 0.1 | 0
  New onset of atrial fibrillation at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  New onset of atrial fibrillation at 1 Year Post-Randomization | 2.4 | 2.4 | 3.4
  New onset of atrial flutter at 1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  New onset of atrial flutter at 1 Year Post-Randomization | 0 | 0.1 | 0

11. Other Pre Specified Outcome: Rate of Acute Kidney Injury (AKI; ≤7 Days Post Index Procedure): Based on the AKIN System Stage 3 (Including Renal Replacement Therapy) or Stage 2
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: Participants will be followed peri- and post-procedure, through 7 days post index procedure.
Population: Intention-To-Treat (ITT): This population includes all subjects who sign an ICF, are enrolled in the trial, and are randomized, whether or not an assigned study device is implanted. A subject treatment group is based on the randomization assignment.
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  Acute kidney injury based on AKIN System Stage 3 (including renal replacement therapy) or Stage 2 | 0 | 0 | 0
  Acute kidney injury based on AKIN System Stage 2 | 0 | 0 | 0
  Acute kidney injury based on AKIN System Stage 3 (including renal replacement therapy) | 0 | 0 | 0

12. Other Pre Specified Outcome: Rate of Coronary Obstruction: Periprocedural
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) - based on VARC endpoints and definitions.
Time Frame: Participants will be followed through 72 hours post index procedure
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants | 0.4 | 0.3 | 0.7

13. Other Pre Specified Outcome: Rate of Ventricular Septal Perforation: Periprocedural
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: Participants will be followed through 72 hours post index procedure
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants | 0.3 | 0.0 | 0.0

14. Other Pre Specified Outcome: Rate of Mitral Apparatus Damage: Periprocedural
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: Participants will be followed through 72 hours post index procedure
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants | 0 | 0 | 0

15. Other Pre Specified Outcome: Rate of Cardiac Tamponade: Periprocedural
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: Participants will be followed through 72 hours post index procedure
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Groups:
- ACURATE neo 2 Valve - Main Randomized: Patients assigned to this group will be implanted with ACURATE neo2™ transfemoral TAVR System.
  *A subset of subjects will also be enrolled in the 4D CT Imaging Substudy.
Arm/Group | ACURATE neo 2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants | 0.4 | 0.3 | 0.7

16. Other Pre Specified Outcome: Rate of Valve Migration
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants
  Discharge/7 Days Post-Randomization (whichever comes first) | 0.1 | 0.3 | 0.0
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 0.1 | 0.3 | 0.0
  6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post-Randomization | 0.1 | 0.3 | 0.0
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 0.1 | 0.3 | 0.0

17. Other Pre Specified Outcome: Rate of Valve Embolization
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants
  Discharge/7 Days Post-Randomization (whichever comes first) | 0.9 | 0.7 | 0.0
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 1.0 | 0.7 | 0.0
  6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post-Randomization | 1.0 | 0.7 | 0.0
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 1.0 | 0.7 | 0.0

18. Other Pre Specified Outcome: Rate of Ectopic Valve Deployment
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: Participants will be followed peri- and post-procedure through discharge or 7 days post-procedure (whichever comes first).
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants | 0.1 | 0.7 | 0.0

19. Other Pre Specified Outcome: Rate of Transcatheter Aortic Valve (TAV)-In-TAV Deployment
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants
  Discharge/7 Days Post- Randomization | 0.7 | 0.1 | 0.0
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 0.7 | 0.1 | 0.0
  6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post-Randomization | 0.7 | 0.1 | 0.7
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 0.7 | 0.1 | 0.7

20. Other Pre Specified Outcome: Rate of Prosthetic Aortic Valve Thrombosis
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants
  Discharge/7 Days Post-Randomization | 0.0 | 0.0 | 0.0
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 0.0 | 0.1 | 0.0
  6 Months Post -Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post -Randomization | 0.4 | 1.8 | 0.0
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 0.7 | 2.6 | 0.0

21. Other Pre Specified Outcome: Rate of Prosthetic Aortic Valve Endocarditis
Description: Safety outcome adjudicated by an independent Clinical Events Committee (CEC) based on VARC-2 endpoints and definitions.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants
  Discharge/7 Days Post-Randomization | 0.0 | 0.0 | 0.0
  30 Days Post-Randomization: number analyzed (Participants) | 734 | 737 | 148
  30 Days Post-Randomization | 0.0 | 0.0 | 0.0
  6 Months Post-Randomization: number analyzed (Participants) | 729 | 731 | 148
  6 Months Post-Randomization | 0.0 | 0.0 | 0.0
  1 Year Post-Randomization: number analyzed (Participants) | 718 | 719 | 146
  1 Year Post-Randomization | 0.1 | 0.1 | 0.0

22. Other Pre Specified Outcome: Rate of Successful Vascular Access, Delivery and Deployment of the Study Valve, and Successful Retrieval of the Delivery System (Site Reported Assessment)
Description: Device Performance outcome, as measured by site reported data based on VARC-2 endpoints and definitions.
Time Frame: Participants will be followed for the duration of their procedure, an expected average of 1 Day (peri- and post-procedure)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants | 98.6 | 99.3 | 100.0

23. Other Pre Specified Outcome: Grade of Aortic Valve Regurgitation: Paravalvular, Central and Combined (Echocardiographic Assessment)
Description: Grade of Aortic Regurgitation as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Time Frame: Participants will be assessed pre-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 Days, 6 Months, and 1 Year. Data for 2-5 years, 7 years, and 10 years will be posted once data is complete.
Population: Intention-To-Treat (ITT): This population includes all subjects who sign an ICF, are enrolled in the trial, and are randomized, whether or not an assigned study device is implanted. A subject treatment group is based on the randomization assignment.
  Number analyzed participants is based on central echo core lab data. Blank data fields or data recorded in the clinical database as 'Not evaluable' are considered missing.
Measure: Number; unit: percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
percentage of participants
  Total aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - None/Trace: number analyzed (Participants) | 721 | 726 | 146
  Total aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - None/Trace | 74.9 | 85.9 | 68.5
  Total aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Mild: number analyzed (Participants) | 721 | 726 | 146
  Total aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Mild | 23.9 | 13.8 | 29.5
  Total aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Moderate: number analyzed (Participants) | 721 | 726 | 146
  Total aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Moderate | 1.1 | 0.3 | 2.1
  Total aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Severe: number analyzed (Participants) | 721 | 726 | 146
  Total aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Severe | 0.1 | 0 | 0
  Central aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - None/Trace: number analyzed (Participants) | 721 | 726 | 146
  Central aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - None/Trace | 98.8 | 99.9 | 97.3
  Central aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Mild: number analyzed (Participants) | 721 | 726 | 146
  Central aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Mild | 1.2 | 0.1 | 2.7
  Central aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Moderate: number analyzed (Participants) | 721 | 726 | 146
  Central aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Moderate | 0 | 0 | 0
  Central aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Severe: number analyzed (Participants) | 721 | 726 | 146
  Central aortic regurgitation (AR) at Discharge/7 Days Post-Procedure - Severe | 0 | 0 | 0
  Aortic paravalvular regurgitation (PVL) at Discharge/7 Days Post-Procedure - None/Trace: number analyzed (Participants) | 721 | 726 | 146
  Aortic paravalvular regurgitation (PVL) at Discharge/7 Days Post-Procedure - None/Trace | 75.9 | 86.1 | 70.5
  Aortic paravalvular regurgitation (PVL) at Discharge/7 Days Post-Procedure - Mild: number analyzed (Participants) | 721 | 726 | 146
  Aortic paravalvular regurgitation (PVL) at Discharge/7 Days Post-Procedure - Mild | 23.0 | 13.6 | 28.1
  Aortic paravalvular regurgitation (PVL) at Discharge/7 Days Post-Procedure - Moderate: number analyzed (Participants) | 721 | 726 | 146
  Aortic paravalvular regurgitation (PVL) at Discharge/7 Days Post-Procedure - Moderate | 1.0 | 0.3 | 1.4
  Aortic paravalvular regurgitation (PVL) at Discharge/7 Days Post-Procedure - Severe: number analyzed (Participants) | 721 | 726 | 146
  Aortic paravalvular regurgitation (PVL) at Discharge/7 Days Post-Procedure - Severe | 0.1 | 0 | 0
  Total aortic regurgitation (AR) at 30 Days Post-Procedure - None/Trace: number analyzed (Participants) | 691 | 695 | 138
  Total aortic regurgitation (AR) at 30 Days Post-Procedure - None/Trace | 57.1 | 75.5 | 52.2
  Total aortic regurgitation (AR) at 30 Days Post-Procedure - Mild: number analyzed (Participants) | 691 | 695 | 138
  Total aortic regurgitation (AR) at 30 Days Post-Procedure - Mild | 38.6 | 23.5 | 44.9
  Total aortic regurgitation (AR) at 30 Days Post-Procedure - Moderate: number analyzed (Participants) | 691 | 695 | 138
  Total aortic regurgitation (AR) at 30 Days Post-Procedure - Moderate | 4.1 | 1.0 | 2.9
  Total aortic regurgitation (AR) at 30 Days Post-Procedure - Severe: number analyzed (Participants) | 691 | 695 | 138
  Total aortic regurgitation (AR) at 30 Days Post-Procedure - Severe | 0.1 | 0 | 0
  Central aortic regurgitation (AR) at 30 Days Post-Procedure - None/Trace: number analyzed (Participants) | 691 | 695 | 138
  Central aortic regurgitation (AR) at 30 Days Post-Procedure - None/Trace | 97.7 | 99.9 | 97.1
  Central aortic regurgitation (AR) at 30 Days Post-Procedure - Mild: number analyzed (Participants) | 691 | 695 | 138
  Central aortic regurgitation (AR) at 30 Days Post-Procedure - Mild | 2.2 | 0.1 | 2.9
  Central aortic regurgitation (AR) at 30 Days Post-Procedure - Moderate: number analyzed (Participants) | 691 | 695 | 138
  Central aortic regurgitation (AR) at 30 Days Post-Procedure - Moderate | 0.1 | 0 | 0
  Central aortic regurgitation (AR) at 30 Days Post-Procedure - Severe: number analyzed (Participants) | 691 | 695 | 138
  Central aortic regurgitation (AR) at 30 Days Post-Procedure - Severe | 0 | 0 | 0
  Aortic paravalvular regurgitation (PVL) at 30 Days Post-Procedure - None/Trace: number analyzed (Participants) | 691 | 695 | 138
  Aortic paravalvular regurgitation (PVL) at 30 Days Post-Procedure - None/Trace | 58.5 | 75.8 | 54.3
  Aortic paravalvular regurgitation (PVL) at 30 Days Post-Procedure - Mild: number analyzed (Participants) | 691 | 695 | 138
  Aortic paravalvular regurgitation (PVL) at 30 Days Post-Procedure - Mild | 38.1 | 23.2 | 42.8
  Aortic paravalvular regurgitation (PVL) at 30 Days Post-Procedure - Moderate: number analyzed (Participants) | 691 | 695 | 138
  Aortic paravalvular regurgitation (PVL) at 30 Days Post-Procedure - Moderate | 3.3 | 1.0 | 2.9
  Aortic paravalvular regurgitation (PVL) at 30 Days Post-Procedure - Severe: number analyzed (Participants) | 691 | 695 | 138
  Aortic paravalvular regurgitation (PVL) at 30 Days Post-Procedure - Severe | 0.1 | 0 | 0
  Total aortic regurgitation (AR) at 6 Months Post-Procedure - None/Trace: number analyzed (Participants) | 612 | 627 | 117
  Total aortic regurgitation (AR) at 6 Months Post-Procedure - None/Trace | 53.0 | 70.1 | 57.3
  Total aortic regurgitation (AR) at 6 Months Post-Procedure - Mild: number analyzed (Participants) | 612 | 627 | 117
  Total aortic regurgitation (AR) at 6 Months Post-Procedure - Mild | 41.8 | 29.2 | 38.5
  Total aortic regurgitation (AR) at 6 Months Post-Procedure - Moderate: number analyzed (Participants) | 612 | 627 | 117
  Total aortic regurgitation (AR) at 6 Months Post-Procedure - Moderate | 5.1 | 0.8 | 4.3
  Total aortic regurgitation (AR) at 6 Months Post-Procedure - Severe: number analyzed (Participants) | 612 | 627 | 117
  Total aortic regurgitation (AR) at 6 Months Post-Procedure - Severe | 0.2 | 0 | 0
  Central aortic regurgitation (AR) at 6 Months Post-Procedure - None/Trace: number analyzed (Participants) | 612 | 627 | 117
  Central aortic regurgitation (AR) at 6 Months Post-Procedure - None/Trace | 96.6 | 99.0 | 96.6
  Central aortic regurgitation (AR) at 6 Months Post-Procedure - Mild: number analyzed (Participants) | 612 | 627 | 117
  Central aortic regurgitation (AR) at 6 Months Post-Procedure - Mild | 3.1 | 1.0 | 3.4
  Central aortic regurgitation (AR) at 6 Months Post-Procedure - Moderate: number analyzed (Participants) | 612 | 627 | 117
  Central aortic regurgitation (AR) at 6 Months Post-Procedure - Moderate | 0.3 | 0 | 0
  Central aortic regurgitation (AR) at 6 Months Post-Procedure - Severe: number analyzed (Participants) | 612 | 627 | 117
  Central aortic regurgitation (AR) at 6 Months Post-Procedure - Severe | 0 | 0 | 0
  Aortic paravalvular regurgitation (PVL) at 6 Months Post-Procedure - None/Trace: number analyzed (Participants) | 612 | 627 | 117
  Aortic paravalvular regurgitation (PVL) at 6 Months Post-Procedure - None/Trace | 54.6 | 71.0 | 58.1
  Aortic paravalvular regurgitation (PVL) at 6 Months Post-Procedure - Mild: number analyzed (Participants) | 612 | 627 | 117
  Aortic paravalvular regurgitation (PVL) at 6 Months Post-Procedure - Mild | 40.8 | 28.2 | 37.6
  Aortic paravalvular regurgitation (PVL) at 6 Months Post-Procedure - Moderate: number analyzed (Participants) | 612 | 627 | 117
  Aortic paravalvular regurgitation (PVL) at 6 Months Post-Procedure - Moderate | 4.4 | 0.8 | 4.3
  Aortic paravalvular regurgitation (PVL) at 6 Months Post-Procedure - Severe: number analyzed (Participants) | 612 | 627 | 117
  Aortic paravalvular regurgitation (PVL) at 6 Months Post-Procedure - Severe | 0.2 | 0 | 0
  Total aortic regurgitation (AR) at 1 Year Post-Procedure - None/Trace: number analyzed (Participants) | 616 | 628 | 123
  Total aortic regurgitation (AR) at 1 Year Post-Procedure - None/Trace | 52.6 | 73.4 | 64.2
  Total aortic regurgitation (AR) at 1 Year Post-Procedure - Mild: number analyzed (Participants) | 616 | 628 | 123
  Total aortic regurgitation (AR) at 1 Year Post-Procedure - Mild | 42.5 | 24.8 | 32.5
  Total aortic regurgitation (AR) at 1 Year Post-Procedure - Moderate: number analyzed (Participants) | 616 | 628 | 123
  Total aortic regurgitation (AR) at 1 Year Post-Procedure - Moderate | 4.4 | 1.8 | 3.3
  Total aortic regurgitation (AR) at 1 Year Post-Procedure - Severe: number analyzed (Participants) | 616 | 628 | 123
  Total aortic regurgitation (AR) at 1 Year Post-Procedure - Severe | 0.5 | 0 | 0
  Central aortic regurgitation (AR) at 1 Year Post-Procedure - None/Trace: number analyzed (Participants) | 616 | 628 | 123
  Central aortic regurgitation (AR) at 1 Year Post-Procedure - None/Trace | 95.0 | 99.4 | 95.9
  Central aortic regurgitation (AR) at 1 Year Post-Procedure - Mild: number analyzed (Participants) | 616 | 628 | 123
  Central aortic regurgitation (AR) at 1 Year Post-Procedure - Mild | 4.7 | 0.6 | 4.1
  Central aortic regurgitation (AR) at 1 Year Post-Procedure - Moderate: number analyzed (Participants) | 616 | 628 | 123
  Central aortic regurgitation (AR) at 1 Year Post-Procedure - Moderate | 0.3 | 0 | 0
  Central aortic regurgitation (AR) at 1 Year Post-Procedure - Severe: number analyzed (Participants) | 616 | 628 | 123
  Central aortic regurgitation (AR) at 1 Year Post-Procedure - Severe | 0 | 0 | 0
  Aortic paravalvular regurgitation (PVL) at 1 Year Post-Procedure - None/Trace: number analyzed (Participants) | 616 | 628 | 123
  Aortic paravalvular regurgitation (PVL) at 1 Year Post-Procedure - None/Trace | 55.5 | 74.0 | 66.7
  Aortic paravalvular regurgitation (PVL) at 1 Year Post-Procedure - Mild: number analyzed (Participants) | 616 | 628 | 123
  Aortic paravalvular regurgitation (PVL) at 1 Year Post-Procedure - Mild | 40.7 | 24.2 | 30.9
  Aortic paravalvular regurgitation (PVL) at 1 Year Post-Procedure - Moderate: number analyzed (Participants) | 616 | 628 | 123
  Aortic paravalvular regurgitation (PVL) at 1 Year Post-Procedure - Moderate | 3.2 | 1.8 | 2.4
  Aortic paravalvular regurgitation (PVL) at 1 Year Post-Procedure - Severe: number analyzed (Participants) | 616 | 628 | 123
  Aortic paravalvular regurgitation (PVL) at 1 Year Post-Procedure - Severe | 0.5 | 0 | 0

24. Other Pre Specified Outcome: Rate of Device Success
Description: Absence of procedural mortality, correct positioning of a single transcatheter valve in the proper anatomical location, and intended performance of the study device (indexed effective orifice area [iEOA] >0.85 cm2/m2 for BMI <30 kg/cm2 and iEOA >0.70 cm2/m2 for BMI ≥30 kg/cm2 plus either a mean aortic valve gradient <20 mmHg or a peak velocity < 3m, and no moderate or severe prosthetic valve aortic regurgitation) based on VARC-2 endpoints and definitions.
Time Frame: Participants will be followed for the duration of their procedure, an expected average of 1 Day (post-procedure)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants
  Device Success | 74.1 | 81.8 | 57.0
  Absence of procedural mortality | 99.6 | 100.0 | 100.0
  Correct positioning of a single valve into the proper anatomical location | 98.4 | 99.1 | 100.0
  Intended performance of the study device | 75.8 | 82.5 | 57.0
  iEOA >0.85 cm2/m2 for BMI <30 kg/m2 and iEOA >0.70 cm2/m2 for BMI ≥30 kg/m2 (AND) | 77.0 | 83.7 | 60.4
  Mean aortic valve gradient <20 mmHg OR peak velocity <3m/sec (AND) | 99.0 | 98.3 | 96.5
  No moderate or severe prosthetic valve aortic regurgitation | 98.8 | 99.7 | 97.9

25. Other Pre Specified Outcome: Effective Orifice Area (EOA)
Description: Effective Orifice Area (EOA), as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Time Frame: as for outcome 23
Population: Intention-To-Treat (ITT): This population includes all subjects who sign an Informed Consent Form, are enrolled in the trial, and are randomized, whether or not an assigned study device is implanted. A subject treatment group is based on the randomization assignment.
  Number analyzed participants is based on central echo core lab data. Blank data fields or data recorded in the clinical database as 'Not evaluable' are considered missing.
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
cm2
  Discharge/7 Days Post-Procedure: number analyzed (Participants) | 652 | 663 | 135
  Discharge/7 Days Post-Procedure | 1.77 (0.3) | 1.82 (032) | 1.68 (0.34)
  30 Days Post-Procedure: number analyzed (Participants) | 645 | 651 | 129
  30 Days Post-Procedure | 1.76 (0.29) | 1.78 (0.31) | 1.65 (0.34)
  6 Months Post-Procedure: number analyzed (Participants) | 576 | 589 | 109
  6 Months Post-Procedure | 1.76 (0.28) | 1.77 (0.31) | 1.65 (0.31)
  1 Year Post-Procedure: number analyzed (Participants) | 573 | 581 | 112
  1 Year Post-Procedure | 1.77 (0.28) | 1.78 (0.30) | 1.64 (0.32)

26. Other Pre Specified Outcome: Mean Aortic Gradient
Description: Mean Aortic Gradient as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Time Frame: as for outcome 23
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
mmHg
  Discharge/7 Days Post-Procedure: number analyzed (Participants) | 704 | 708 | 142
  Discharge/7 Days Post-Procedure | 9.0 (3.9) | 10.2 (4.2) | 10.0 (4.7)
  30 Days Post-Procedure: number analyzed (Participants) | 679 | 685 | 133
  30 Days Post-Procedure | 8 (3.2) | 10.1 (4.7) | 8.1 (3.3)
  6 Months Post-Procedure: number analyzed (Participants) | 604 | 616 | 115
  6 Months Post-Procedure | 8.1 (3.3) | 10.6 (5.1) | 8.1 (4.0)
  1 Year Post-Procedure: number analyzed (Participants) | 604 | 615 | 120
  1 Year Post-Procedure | 7.9 (3.3) | 10.7 (5.0) | 8.4 (3.4)

27. Other Pre Specified Outcome: New York Heart Association (NYHA) Functional Status Classification
Description: Health status evaluated by New York Heart Association (NYHA) Classification.
  NYHA Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Time Frame: Participants will be followed peri- and post-procedure, at discharge or 7 days post-procedure (whichever comes first), 30 Days, 6 Months, and 1 Year. Data for 2-5 years, 7 years, and 10 years will be posted once data is complete.
Population: Intention-To-Treat (ITT): This population includes all subjects who sign an Informed Consent Form, are enrolled in the trial, and are randomized, whether or not an assigned study device is implanted. A subject treatment group is based on the randomization assignment.
  NYHA class denominator is the number of subjects with non-missing NYHA class at the studied timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Percentage of participants
  Discharge/7 Days Post Procedure NYHA Functional Class - I: number analyzed (Participants) | 715 | 716 | 147
  Discharge/7 Days Post Procedure NYHA Functional Class - I | 34.1 | 32.0 | 32.7
  Discharge/7 Days Post-Procedure NYHA Functional Class - II: number analyzed (Participants) | 715 | 716 | 147
  Discharge/7 Days Post-Procedure NYHA Functional Class - II | 49.4 | 52.4 | 49.0
  Discharge/7 Days Post-Procedure NYHA Functional Class - III: number analyzed (Participants) | 715 | 716 | 147
  Discharge/7 Days Post-Procedure NYHA Functional Class - III | 15.8 | 15.5 | 18.4
  Discharge/7 Days Post-Procedure NYHA Functional Class - IV: number analyzed (Participants) | 715 | 716 | 147
  Discharge/7 Days Post-Procedure NYHA Functional Class - IV | 0.7 | 0.1 | 0.0
  30 Days Post-Procedure NYHA Functional Class - I: number analyzed (Participants) | 699 | 694 | 145
  30 Days Post-Procedure NYHA Functional Class - I | 57.7 | 60.1 | 57.2
  30 Days Post-Procedure NYHA Functional Class - II: number analyzed (Participants) | 699 | 694 | 145
  30 Days Post-Procedure NYHA Functional Class - II | 37.8 | 35.0 | 39.3
  30 Days Post-Procedure NYHA Functional Class - III: number analyzed (Participants) | 699 | 694 | 145
  30 Days Post-Procedure NYHA Functional Class - III | 4.3 | 4.9 | 3.4
  30 Days Post-Procedure NYHA Functional Class - IV: number analyzed (Participants) | 699 | 694 | 145
  30 Days Post-Procedure NYHA Functional Class - IV | 0.3 | 0.0 | 0.0
  6 Months Post-Procedure NYHA Functional Class - I: number analyzed (Participants) | 633 | 634 | 132
  6 Months Post-Procedure NYHA Functional Class - I | 65.1 | 66.2 | 64.4
  6 Months Post-Procedure NYHA Functional Class - II: number analyzed (Participants) | 633 | 634 | 132
  6 Months Post-Procedure NYHA Functional Class - II | 29.9 | 29.3 | 31.1
  6 Months Post-Procedure NYHA Functional Class - III: number analyzed (Participants) | 633 | 634 | 132
  6 Months Post-Procedure NYHA Functional Class - III | 4.6 | 4.4 | 4.5
  6 Months Post-Procedure NYHA Functional Class - IV: number analyzed (Participants) | 633 | 634 | 132
  6 Months Post-Procedure NYHA Functional Class - IV | 0.5 | 0.0 | 0.0
  1 Year Post-Procedure NYHA Functional Class - I: number analyzed (Participants) | 630 | 630 | 126
  1 Year Post-Procedure NYHA Functional Class - I | 64.9 | 64.4 | 60.3
  1 Year Post-Procedure NYHA Functional Class - II: number analyzed (Participants) | 630 | 630 | 126
  1 Year Post-Procedure NYHA Functional Class - II | 31.9 | 31.1 | 35.7
  1 Year Post-Procedure NYHA Functional Class - III: number analyzed (Participants) | 630 | 630 | 126
  1 Year Post-Procedure NYHA Functional Class - III | 3.0 | 4.4 | 4.0
  1 Year Post-Procedure NYHA Functional Class - IV: number analyzed (Participants) | 630 | 630 | 126
  1 Year Post-Procedure NYHA Functional Class - IV | 0.2 | 0.0 | 0.0

28. Other Pre Specified Outcome: Health Status: Kansas City Cardiomyopathy Questionnaire (KCCQ) Quality of Life Assessment - Change From Baseline
Description: Health Status additional outcome KCCQ Analysis - Overall Summary Score change from Baseline.
  Kansas City Cardiomyopathy Questionnaire (KCCQ): Quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  Overall Summary Score - mean of score 1, 5, 7, and 8
Time Frame: Participants will be assessed at baseline, 30 Days, and 1 Year. Data for 5 years will be posted once data is complete.
Population: Intention-To-Treat (ITT): This population includes all subjects who sign an Informed Consent Form, are enrolled in the trial, and are randomized, whether or not an assigned study device is implanted. A subject treatment group is based on the randomization assignment.
  Note: paired analysis includes subjects with non-missing data at both baseline and the specific follow-up visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Score on a scale
  Baseline - Overall Summary Score: number analyzed (Participants) | 737 | 739 | 144
  Baseline - Overall Summary Score | 62.4 (22.3) | 62.2 (21.9) | 62.0 (21.5)
  Change from Baseline to 30 Days - Overall Summary Score: number analyzed (Participants) | 700 | 701 | 140
  Change from Baseline to 30 Days - Overall Summary Score | 18.1 (21.6) | 17.8 (22.1) | 19.8 (21.1)
  Change from Baseline to 1 Year - Overall Summary Score: number analyzed (Participants) | 631 | 628 | 126
  Change from Baseline to 1 Year - Overall Summary Score | 19.4 (22.2) | 20.0 (22.1) | 19.8 (20.8)

29. Other Pre Specified Outcome: Health Status: SF-12 Quality of Life Questionnaire Assessment - Change From Baseline
Description: Health Status outcome - SF-12 - Baseline scores and changes from Baseline at 30 Days and 1 Year.
  12 Item Short Form Health Survey (SF-12): Measures functional health and well-being. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Participants will be assessed at baseline, 30 Days, and 1 Year. Data for 5 years will be posted once data is complete.
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
Number analyzed (Participants) | 752 | 748 | 148
Score on a scale
  Baseline - Physical Summary Score: number analyzed (Participants) | 732 | 735 | 144
  Baseline - Physical Summary Score | 36.9 (10.7) | 36.1 (11.0) | 36.4 (10.2)
  Baseline - Mental Health Summary Score: number analyzed (Participants) | 732 | 735 | 144
  Baseline - Mental Health Summary Score | 51.7 (10.0) | 51.8 (10.3) | 51.6 (9.1)
  Change from Baseline to 30 Days - Physical Summary Score: number analyzed (Participants) | 690 | 691 | 139
  Change from Baseline to 30 Days - Physical Summary Score | 4.8 (9.9) | 5.4 (10.5) | 5.7 (10.6)
  Change from Baseline to 30 Days - Mental Health Summary Score: number analyzed (Participants) | 690 | 691 | 139
  Change from Baseline to 30 Days - Mental Health Summary Score | 2.8 (11.1) | 2.3 (11.1) | 3.2 (10.7)
  Change from Baseline to 1 Year - Physical Summary Score: number analyzed (Participants) | 626 | 622 | 125
  Change from Baseline to 1 Year - Physical Summary Score | 5.2 (11.0) | 5.4 (11.5) | 4.8 (10.2)
  Change from Baseline to 1 Year - Mental Health Summary Score: number analyzed (Participants) | 626 | 622 | 125
  Change from Baseline to 1 Year - Mental Health Summary Score | 2.0 (10.8) | 2.1 (11.1) | 1.6 (10.4)

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Event reporting is required from randomization for the Main Randomized cohort and from index procedure for the Roll-in cohort. SAEs are reported by the sites through the end of study while AEs are reported through 1-year post-procedure.
  Events are reported for the ITT population.
Groups:
- Commercial Valve - Main Randomized: Medtronic CoreValve TAVR System OR, Edwards SAPIEN 3 TAVR System.
  Patients assigned to this group will be implanted with commercially available balloon-expandable SAPIEN 3™ Transcatheter Heart Valve or future iteration (SAPIEN 3; Edwards Lifesciences LLC, Irvine, CA, USA) or a commercially available self-expanding CoreValve® Transcatheter Aortic Valve Replacement System, CoreValve® Evolut™ R Recapturable TAVR System, EVOLUT™ PRO System, or future iteration (CoreValve; Medtronic, Inc., Dublin, Ireland) TAVR device.
  *A minimum of 200 subjects will also be enrolled in the 4D CT Imaging Substudy.
Arm/Group | ACURATE neo2 Valve - Main Randomized | Commercial Valve - Main Randomized | ACURATE neo2 Valve - Single-arm Roll-in
All-Cause Mortality (participants affected / at risk) | 36/752 | 28/748 | 7/148
Serious Adverse Events (participants affected / at risk) | 389/752 | 381/748 | 81/148
Other Adverse Events (participants affected / at risk) | 155/752 | 145/748 | 26/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACURATE neo2 Valve - Main Randomized (N=752) | Commercial Valve - Main Randomized (N=748) | ACURATE neo2 Valve - Single-arm Roll-in (N=148)
Anaemia (Blood and lymphatic system disorders) | 10 (10) | 4 (4) | 4 (5)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 12 (13) | 4 (4) | 1 (2)
Acute myocardial infarction (Cardiac disorders) | 13 (13) | 5 (6) | 0 (0)
Angina pectoris (Cardiac disorders) | 3 (3) | 5 (5) | 0 (0)
Angina unstable (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Aortic valve thickening (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriospasm coronary (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 32 (37) | 38 (40) | 7 (11)
Atrial flutter (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 3 (3) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 52 (53) | 68 (70) | 7 (7)
Atrioventricular block first degree (Cardiac disorders) | 5 (5) | 7 (7) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 7 (7) | 6 (6) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4) | 9 (9) | 0 (0)
Bundle branch block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 32 (32) | 30 (30) | 2 (2)
Bundle branch block right (Cardiac disorders) | 2 (2) | 5 (5) | 0 (0)
Cardiac arrest (Cardiac disorders) | 11 (11) | 3 (3) | 2 (2)
Cardiac failure (Cardiac disorders) | 7 (8) | 8 (9) | 1 (2)
Cardiac failure acute (Cardiac disorders) | 9 (10) | 8 (8) | 3 (4)
Cardiac failure congestive (Cardiac disorders) | 22 (28) | 19 (22) | 8 (11)
Cardiac perforation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 4 (4) | 0 (0)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Coronary artery thrombosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperdynamic left ventricle (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Low cardiac output syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 5 (5) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 7 (7) | 2 (3) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 3 (4) | 3 (3) | 0 (0)
Myocardial rupture (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Nodal rhythm (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Paravalvular aortic regurgitation (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Prosthetic cardiac valve thrombosis (Cardiac disorders) | 0 (0) | 6 (6) | 0 (0)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 4 (4) | 7 (7) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 2 (3) | 5 (5) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (3) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 4 (4) | 3 (3) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Skin malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 2 (2) | 1 (2)
Cataract nuclear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Retinal infarction (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal strangulated hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 (7) | 8 (10) | 1 (1)
Gastrointestinal vascular malformation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Internal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (2) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oesophageal food impaction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (3) | 1 (1) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Asthenia (General disorders) | 3 (3) | 2 (2) | 0 (0)
Catheter site haematoma (General disorders) | 3 (3) | 3 (3) | 1 (1)
Catheter site haemorrhage (General disorders) | 4 (4) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 2 (2) | 0 (0) | 0 (0)
Cyst (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 11 (11) | 4 (4) | 0 (0)
Device embolisation (General disorders) | 7 (7) | 4 (4) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 2 (2) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0) | 0 (0)
Abdominal wall infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 4 (4) | 3 (3) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 7 (7) | 2 (2) | 5 (5)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Clostridial sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 12 (12) | 7 (7) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Endocarditis (Infections and infestations) | 2 (2) | 2 (3) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Necrotising soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (16) | 19 (19) | 5 (5)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 9 (9) | 14 (16) | 5 (5)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic encephalopathy (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 2 (2) | 3 (3) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 17 (19) | 10 (10) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 5 (5) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Device deployment issue (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 11 (11) | 6 (6) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Structural valve deterioration (Injury, poisoning and procedural complications) | 0 (0) | 6 (6) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Trunk injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Urethral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Vascular access site complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular procedure complication (Injury, poisoning and procedural complications) | 4 (5) | 3 (3) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 4 (4) | 4 (4) | 3 (3)
Vascular pseudoaneurysm thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bleeding time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
CSF test abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Echocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lactescent serum (Investigations) | 0 (0) | 1 (1) | 0 (0)
Pedal pulse decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 2 (2) | 2 (2) | 2 (2)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 3 (3) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (7) | 6 (6) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acute megakaryocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5) | 2 (2) | 0 (0)
Benign uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 4 (4) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Cerebellar ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (5) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 3 (3) | 2 (2)
Cerebral microhaemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 28 (30) | 12 (12) | 6 (6)
Chorea (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 5 (5) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 6 (6) | 4 (4) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Periventricular leukomalacia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 8 (8) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 8 (9) | 5 (5) | 6 (6)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 12 (13) | 7 (7) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 1 (1) | 0 (0)
Device failure (Product Issues) | 3 (3) | 0 (0) | 0 (0)
Device leakage (Product Issues) | 3 (3) | 2 (2) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
Delirium tremens (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 4 (4) | 6 (6) | 1 (1)
Substance abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 22 (26) | 17 (18) | 7 (8)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (6) | 6 (7) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (4) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 3 (3) | 3 (3) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 2 (2) | 1 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (3) | 2 (3)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 2 (2)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 17 (18) | 2 (2)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Air embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (4) | 4 (4) | 0 (0)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral artery dissection (Vascular disorders) | 2 (2) | 3 (3) | 0 (0)
Haematoma (Vascular disorders) | 3 (3) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 6 (6) | 2 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 4 (4) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 15 (15) | 6 (6) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Iliac artery perforation (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphorrhoea (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Necrosis ischaemic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Paradoxical embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Penetrating aortic ulcer (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 3 (3) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery dissection (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 2 (2) | 3 (3) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 6 (6) | 2 (2) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 2 (2) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subclavian artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subclavian artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Vascular calcification (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACURATE neo2 Valve - Main Randomized (N=752) | Commercial Valve - Main Randomized (N=748) | ACURATE neo2 Valve - Single-arm Roll-in (N=148)
Atrioventricular block first degree (Cardiac disorders) | 49 (50) | 48 (48) | 9 (9)
Bundle branch block left (Cardiac disorders) | 121 (122) | 111 (114) | 13 (13)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 8 (8) — and Administration site conditions

LIMITATIONS AND CAVEATS:
Trial-related factors

* First RCT experience with ACURATE neo2 enrolled patients of all risks
* Control arm included two comparator devices, with operator selection of preferred Control at time of randomization

Enrollment factors

* COVID - impact on staffing resources (hospital & sponsor support); supply constraints; investigational cases deprioritized relative to commercial cases
* Operators less experienced with ACURATE neo2 compared to Control devices

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A contractual agreement is in place between the PIs and the Sponsor that restricts the rights to discuss or publish trial results without prior review by the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT03735667/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT03735667/SAP_002.pdf